CLINICAL TRIAL: NCT02586961
Title: Nebulized Adrenalin and Oral Betamethasone in Children With Bronchiolitis Attending Pediatric Emergencies : a Multicentre Randomized Controlled Trial
Brief Title: Nebulized Adrenalin and Oral Betamethasone in Children With Bronchiolitis Attending Pediatric Emergencies.
Acronym: EPIDEX
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Removal of Adrénaline lots for safety reasons.
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P140929; 2015-002477-38 (EudraCT Number)
Record Dates: First submitted 2015-10-18; First posted 2015-10-27 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2016-10

CONDITIONS: Children; Bronchiolitis
Keywords: randomized prospective study; complication rate; bronchiolitis; children
MeSH Terms: conditions — Bronchiolitis | interventions — Saline Solution; Epinephrine; Betamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.9% saline solution - oral betamethasone placebo (Placebo Comparator): Control arm: 0.9% saline solution - oral betamethasone placebo
  Interventions: Drug: 0.9% saline solution; Drug: oral betamethasone placebo
- adrenaline - oral betamethasone (Experimental): Experimental arm : adrenaline and betamethasone
  Interventions: Drug: adrenaline; Drug: oral betamethasone

INTERVENTIONS:
Drug: 0.9% saline solution — Placebo:
  Nebulized 0.9% saline solution
  Arms: 0.9% saline solution - oral betamethasone placebo
Drug: oral betamethasone placebo — placebo of oral betamethasone: equivalent of 1 mg/kg at inclusion followed by five once-daily doses
  Arms: 0.9% saline solution - oral betamethasone placebo
Drug: adrenaline — Catecholamine nebulized adrenaline (3 ml of 1:1000 solution)
  Arms: adrenaline - oral betamethasone
Drug: oral betamethasone — Mineralocorticoid: a short course of oral betamethasone: 1.0 mg/kg at inclusion, followed by five once-daily doses (0.6 mg/kg)
  Arms: adrenaline - oral betamethasone

SUMMARY:
The combined administration of high dose of oral betamethasone and nebulization of adrenaline seems to be an attractive therapeutic alternative for reducing the rate of hospitalization for acute bronchiolitis treated in the emergency department. However, it is essential to confirm the trend previously observed with this treatment before using it in current practice.

DETAILED DESCRIPTION:
Rationale: In infancy, bronchiolitis is the most common acute infection of the lower respiratory tract and is most often caused by the respiratory syncytial virus (RSV). The current treatment of bronchiolitis is controversial. Although meta-analysis of nebulized bronchodilators or corticosteroids treatments failed to show any consistent benefits on admission rate, they remain widely used in pediatric emergency wards. A recent randomized, double-blind, placebo-controlled, clinical trial with a factorial design was conducted to determine whether treatment with nebulized epinephrine, a short course of high dose of oral Betamethasone, or both, resulted in a clinically important decrease in hospital admissions among infants with bronchiolitis who were seen in the emergency department. This study showed that infants in the epinephrine-betamethasone group were significantly less likely than those in the placebo group to be admitted by day 7 (relative risk, 0.65; 95% confidence interval, 0.45 to 0.95, P = 0.02). However, after adjustment for multiple comparisons, this result became insignificant (P = 0.07). This synergistic interaction was not anticipated but gave hope that the association nebulized epinephrine - short course of oral high dose of betamethasone might reduce the risk of hospitalization for infants who consulted pediatric emergencies for a moderate to severe acute bronchiolitis. It is therefore required to conduct a trial dedicated to this evaluation in the French population.

Hypothesis: using Epinephrine-Betamethasone allows to reduce the rate of hospitalization of mild-to-severe acute viral bronchiolitis seen in pediatric emergency departments.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 6 weeks to 12 months admitted in paediatric emergency
* First episode of acute bronchiolitis defined as: expiratory dyspnea with breath slowing and/or sibilants and/or crackles preceded by (or associated with) a nasopharyngitis more or less febrile
* Respiratory distress assessment index score (RDAI) of 4 to 15 after a nasopharyngeal clearance
* Agreement of at least one of the parents for his child to participate in biomedical research
* Affiliation to social security (beneficiary or entitled), except beneficiary of State medical help

Exclusion Criteria:

* Prematurity (less than 37 weeks of gestation)
* Antecedent of invasive respiratory ventilation during neonatal period
* Antecedent of lung or chronic cardiac pathology of wich rhythm disorder, acute obstructive cardiomyopathy and coronary insufficiency
* Immune deficiency
* Active viral infection (hepatitis, zona, herpes, varicella, HIV)
* Proven or suspected tuberculosis
* Exposure to varicella during 15 days before inclusion
* Severe distress (defined as one of following signs: a pulse rate >200/min, respiratory rate >80/min, RDAI score >15, neurological disorders)
* Nebulization (aerosol spray) of Salbutamol or other bronchodilator treatment during the 24 hours before the inclusion
* Inhalation (spray) of Salbutamol during the preceding 24 hours
* Oral or inhaled corticosteroids during the preceding 2 weeks
* Previous episode of wheezing or ascertained diagnosis of asthma
* Hypersensitivity to one of the constituting of oral betamethasone
* Vaccination by living vaccine during the preceding 2 weeks

Ages: 6 Weeks to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 195 (Actual)
Dates: Start 2015-10; Primary Completion 2017-09 (Actual); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Hospital admission up to 7 days after enrollment, which occurred during the visit in the emergency department | 7 days after enrollment
  determine whether treatment with nebulized adrenaline (3 ml of 1:1000 solution) and a short course of oral dexamethasone (1.0 mg/kg) followed by five once-daily doses (0.6 mg/kg) results in a 10% decrease in hospital admissions among infants with mild-to-severe bronchiolitis seen in emergency departments

SECONDARY OUTCOMES:
PICU admission rate following examination in the emergency ward | during the 7 days after enrollment
  Estimate and compare the percentages of infants in each group requiring Pediatric Intensive Care Unit (PICU admission).
Length of hospitalization for infants admitted for bronchiolitis in the following 7 days after inclusion | 7 days after enrollment
  Assess whether experimental treatment reduces healing time and duration of hospitalization of infants included in the study and who have been admitted
Variation of RDAI scores before and after nebulization | between enrollment and an average of 7 days (the end hospitalization)
  Compare clinical scores of respiratory distress before/after treatment
Adverse events during the following 7 days after inclusion | 7 days after enrollment
  Evaluate the tolerance of experimental treatment

CONTACTS AND LOCATIONS:
Overall Officials: Vincent GAJDOS, Principal Investigator — AP-HP, Antoine Béclère Hospital
Locations (1):
- AP-HP, Antoine Béclère Hospital, Clamart, France